CLINICAL TRIAL: NCT06094244
Title: Statins and 90-day Functional Efficiency and Survival in Patients With Spontaneous Intracerebral Hemorrhage
Brief Title: Statins in Patients With Spontaneous Intracerebral Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Karolina Zaryczańska, Karolina Zaryczańska, MD, PhD, Pomeranian Medical University Szczecin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pomeranian MU Szczecin
Record Dates: First submitted 2023-07-19; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Intracerebral Hemorrhage
Keywords: SICH; Spontaneous intracerebral hemorrhage; Statins; Functional efficiency; NIHSS Scale; Rankin Scale; Barthel Scale; Intracerebral Hemorrhage; Stroke
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group I Patients who were not taking statins prior to the occurrence of SICH (Experimental): Patients who were not taking statins prior to the occurrence of SICH.
  Interventions: Other: No drugs
- Group II Patients who were taking statins prior to the occurrence of SICH (Experimental): Patients who were taking statins prior to the occurrence of SICH.
  Interventions: Drug: Atorvastatin; Drug: Rosuvastatin
- Subgroup Ia Patients were not diagnosed to dyslipidemia. They did not receive statins. (Experimental): Patients who were not diagnosed to have dyslipidemia during hospitalization. They did not receive statins.
  Interventions: Other: No drugs
- Subgroup Ib Patients with dyslipidemia Received statins, recommended to take medicine for 90 days. (Experimental): Patients with dyslipidemia diagnosed during hospitalization who received statins and were recommended to take this medicine for 90 days since they occurrence of SICH.
  Interventions: Drug: Atorvastatin; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Atorvastatin — Doses of atorvastatin of up to 20 mg/d.
  Arms: Group II Patients who were taking statins prior to the occurrence of SICH; Subgroup Ib Patients with dyslipidemia Received statins, recommended to take medicine for 90 days.
Drug: Rosuvastatin — Doses of rosuvastatin of up to 10 mg/d.
  Arms: Group II Patients who were taking statins prior to the occurrence of SICH; Subgroup Ib Patients with dyslipidemia Received statins, recommended to take medicine for 90 days.
Other: No drugs — No drugs
  Arms: Group I Patients who were not taking statins prior to the occurrence of SICH; Subgroup Ia Patients were not diagnosed to dyslipidemia. They did not receive statins.

SUMMARY:
The relation between improvement in results of treating spontaneous intracerebral hemorrhage (SICH) and the application of statins has been subject to numerous analyses, and yet still remains debatable. The options of treating SICH are limited, therefore neuroprotective effects of statins have become the subject of interest.

The purpose of this work is to determine whether:

1. the use of statins in the period prior to the spontaneous intracerebral hemorrhage has any impact on the initial neurological condition and the initial radiology
2. continuing the statin treatment commenced before the spontaneous intracerebral hemorrhage or including statins into treatment at the acute stage of the disease deteriorates the course of the disease and prognosis during the in-hospital period
3. continuing treatment with statins after the in-hospital treatment impacts functional efficiency and survival rate within the period of up to 90 days from the symptoms of spontaneous intracerebral hemorrhage occurring.

The prospective study included 153 patients with diagnosed SICH who met the criteria for inclusion based on data collected in the course of interviews, neurological examinations, neuroimaging (head scans or magnetic resonance of the head) and laboratory test results, which additionally made it possible to exclude secondary hemorrhage causes.

During the first stage of the study, patients were assigned to group I (without statins) and group II (taking statins).

During the second stage of the study, having marked the lipid profile within the first three days of stay in hospital and excluded or confirmed dyslipidemia, group I was further divided into subgroups Ia and Ib. Subgroup Ia comprised those who were not diagnosed to have dyslipidemia - they did not receive statins; subgroup Ib comprised those with dyslipidemia who received statins and were recommended to take this medicine for 90 days since they occurrence of SICH. Group II patients continued to take the same dose of statins they had been taking before (atorvastatin or rosuvastatin) or if it had initially been low - increased doses of atorvastatin of up to 20 mg/d and rosuvastatin of up to 10 mg/d. Persons who had never taken that medicine before (subgroup Ib) were administered atorvastatin of 20 mg/day with the recommendation to take it for at least 90 days since the occurrence of SICH symptoms. The analysis pertained to the impact of statins during the acute period of SICH on its in-hospital course.

The third stage consisted in analyzing the condition of the patients post hospitalization with the NIHSS Scale, Barthel Scale and modified Rankin Scale, with an examination carried out on the day they were released from hospital and 90 days from the occurrence of the symptoms of the disease.

The fourth stage consisted in analyzing the survival rate of the patients.

DETAILED DESCRIPTION:
The relation between improvement in results of treating spontaneous intracerebral hemorrhage (SICH) and the application of statins has been subject to numerous analyses, and yet still remains debatable. The options of treating SICH are limited and focus on containing arterial hypertension, treating cerebral edema and providing supportive care, primarily physical and speech therapy, as well as preventing complications in bed-ridden patients in grave medical condition. Therefore, neuroprotective effects of statins have become the subject of interest, especially in the case of diseases with low possibilities of treatment but catastrophic health and social consequences, caused by SICH.

The intended purpose of this work is to determine whether:

1. the use of statins in the period prior to the spontaneous intracerebral hemorrhage has any impact on the initial neurological condition and the initial radiology
2. continuing the statin treatment commenced before the spontaneous intracerebral hemorrhage or including statins into treatment at the acute stage of the disease deteriorates the course of the disease and prognosis during the in-hospital period
3. continuing treatment with statins after the in-hospital treatment impacts functional efficiency and survival rate within the period of up to 90 days from the symptoms of spontaneous intracerebral hemorrhage occurring.

The prospective study included 153 patients with diagnosed SICH who met the criteria for inclusion based on data collected in the course of interviews, neurological examinations, neuroimaging (head scans or magnetic resonance of the head) and laboratory test results, which additionally made it possible to exclude secondary hemorrhage causes.

During the first stage of the study, patients were assigned to group I (without statins) and group II (taking statins).

During the second stage of the study, having marked the lipid profile within the first three days of stay in hospital and excluded or confirmed dyslipidemia, group I was further divided into subgroups Ia and Ib. Subgroup Ia comprised those who were not diagnosed to have dyslipidemia - they did not receive statins; subgroup Ib comprised those with dyslipidemia who received statins and were recommended to take this medicine for 90 days since they occurrence of SICH. Group II patients continued to take the same dose of statins they had been taking before (atorvastatin or rosuvastatin) or if it had initially been low - increased doses of atorvastatin of up to 20 mg/d and rosuvastatin of up to 10 mg/d. Persons who had never taken that medicine before (subgroup Ib) were administered atorvastatin of 20 mg/day with the recommendation to take it for at least 90 days since the occurrence of SICH symptoms. The analysis pertained to the impact of statins during the acute period of SICH on its in-hospital course.

The third stage consisted in analyzing the condition of the patients post hospitalization with the NIHSS Scale, Barthel Scale and modified Rankin Scale, with an examination carried out on the day they were released from hospital and 90 days from the occurrence of the symptoms of the disease. The examination was conducted directly or through a phone conversation with the patient or their caretaker with a uniform set of questions based on a scale.

The fourth stage consisted in analyzing the survival rate of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old
2. Spontaneous intracerebral hemorrhage confirmed by computed tomography/MRI of the head
3. Taking statins: rosuvastatin or atorvastatin for at least 6 months - applies only to group II

Exclusion Criteria:

1. Secondary central nervous system bleeding (e.g. tumor, vascular malformation, haemorrhaged ischemic stroke, coagulopathy, anticoagulant therapy)
2. SAH/traumatic bleeding
3. Accompanying ischemic focus in the brain
4. Infection with fever and/or high inflammatory parameters on the day of admission to the hospital
5. Age under 18 years old

Ages: 36 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
NIHSS | 24 hours
  NIHSS - Assessment of neurological deficit on a scale from 0 to 42. The higher the number, the deeper the neurological deficit.
NIHSS | During hospital stay (up to 14 days)
  NIHSS - Assessment of neurological deficit on a scale from 0 to 42. The higher the number, the deeper the neurological deficit.
Modified Rankin Scale | During hospital stay (up to 14 days)
  Modified Rankin Scale - Assessment of global disability, score range from 0 to 6, where 0 means full disability, 5 means full disability, and 6 means death.
Barthel Scale | During hospital stay (up to 14 days)
  Barthel Scale - Assessment of the deficit in self-care, score from 0 to 100. From 0-20 are patients requiring complete care. 100 points means a person functioning independently.
Mortality | During hospital stay (up to 14 days)
  Mortality Assessment - The number of deaths in a population during a given time or place.
NIHSS | Up to 90 days
  NIHSS - Assessment of neurological deficit on a scale from 0 to 42. The higher the number, the deeper the neurological deficit.
Modified Rankin Scale | Up to 90 days
  Modified Rankin Scale - Assessment of global disability, score range from 0 to 6, where 0 means full disability, 5 means full disability, and 6 means death.
Barthel Scale | Up to 90 days
  Barthel Scale - Assessment of the deficit in self-care, score from 0 to 100. From 0-20 are patients requiring complete care. 100 points means a person functioning independently.
Mortality | Up to 90 days
  Mortality Assessment - The number of deaths in a population during a given time or place.

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Zaryczańska, PhD, MD, Principal Investigator — Pomeranian Medical University
Locations (1):
- Pomeranian Medical University, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No